CLINICAL TRIAL: NCT06215313
Title: EMDR Versus Imagery Rescripting as a Treatment for Trauma-Related Intrusive Images
Brief Title: EMDR Versus Imagery Rescripting for Trauma-Related Intrusions
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Geestelijke Gezondheidszorg Eindhoven (GGzE) (Other)
Collaborators: Maastricht University (Other)
Responsible Party: Principal Investigator, Justine De Rous, junior onderzoeker, Geestelijke Gezondheidszorg Eindhoven (GGzE)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL85848.068.23
Record Dates: First submitted 2023-12-14; First posted 2024-01-22 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Stress Disorders, Post-Traumatic; Depression
Keywords: EMDR; Imagery Rescripting; Personalised treatment; Working mechanisms; Intrusions; PTSD; Depression
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression | interventions — Eye Movement Desensitization Reprocessing

STUDY DESIGN:
Intervention Model Description: This study will use a single-case experimental design (SCED). In this study, there are three groups (PTSD, depression, and PTSD with comorbid depression) and two interventions (EMDR and IR), that is 3 x 2 = 6 simultaneous SCEDs. Seven patients per SCED will be included, i.e., a total of 42 patients. Patients will be randomly assigned to one of the two interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients with PTSD (Experimental): Patients with PTSD will be randomly assigned to either EMDR or IR. They will receive two 75-minute sessions of either EMDR or IR each week, with one additional coaching session in both conditions (EMDR and IR).
  Interventions: Behavioral: Eye Movement Desensitization and Reprocessing; Behavioral: Imagery Rescripting
- Patients with depression (Experimental): Patients with depression will be randomly assigned to either EMDR or IR. They will receive two 75-minute sessions of either EMDR or IR each week, with one additional coaching session in both conditions (EMDR and IR).
  Interventions: Behavioral: Eye Movement Desensitization and Reprocessing; Behavioral: Imagery Rescripting
- Patients with PTSD and depression (Experimental): Patients with PTSD and depression will be randomly assigned to either EMDR or IR. They will receive two 75-minute sessions of either EMDR or IR each week, with one additional coaching session in both conditions (EMDR and IR).
  Interventions: Behavioral: Eye Movement Desensitization and Reprocessing; Behavioral: Imagery Rescripting

INTERVENTIONS:
Behavioral: Eye Movement Desensitization and Reprocessing — In the EMDR condition, the Dutch version of the treatment protocol based on Shapiro's original work (2001) is followed. In the first session, the rationale of EMDR is explained. The patient describes the memory, and identifies the most aversive still image, the associated negative cognition, desired positive cognition, feelings, somatic sensations, and perceived tension, as measured by Subjective Unit of Distress (SUDs). Desensitization then begins by asking patients to focus on the still image while following the movement of a light bar or the therapist's fingers with their eyes (i.e., eye tracking task). Then, in the installation phase, the patient focuses on the positive cognition during the eye tracking task. When the validity of the positive cognition is 6 to 7 on a 7-point Likert scale, a body scan is performed to ensure that no unresolved traumatic material remains. Each session ends with a reflection and debriefing.
  Other Names: EMDR
Behavioral: Imagery Rescripting — The IR condition, following Arntz and Weertman's (1999) protocol, addresses traumatic or aversive memories by creating alternative scenarios. In the first session, the method is explained. The patient describes their memory in the present tense, from the first-person perspective, and describes associated feelings, thoughts, and emotional needs. The therapist then seeks permission to 'enter' the scene, guiding the patient to visualise an alternative, emotionally satisfying course of events. This may involve the therapist or patient intervening in the situation, ensuring the patient's emotional needs are met. The patient then relives the memory from the point of view of their younger self, with the adult-self intervening in the scene. The process continues until all emotional needs are fulfilled. Generally, one trauma memory is rescripted per session. The initial IR session involves therapist-led rescripting, with subsequent sessions encouraging patient-led rescripting whenever possible.
  Other Names: IR

SUMMARY:
The goal of this clinical trial is to investigate the effectiveness and mechanisms of action of trauma treatments in a sample of patients meeting criteria for posttraumatic stress disorder (PTSD), unipolar depression, or both disorders. The main questions it aims to answer are:

* which first line treatment (Eye Movement Desensitization and Reprocessing [EMDR] vs. Imaginary Rescripting [IR]) works better for intrusive experiences in patients with PTSD, patients with a depression, and patients who meet criteria for both diagnoses.
* which mechanisms of action cause the treatment effects.

Participants will

* be randomly assigned to a standard treatment of EMDR or IR
* complete daily questionnaires measuring the outcome measures two weeks before the start of their treatment, during their EMDR or IR treatment, and for one month after their treatment.
* complete questionnaires measuring the outcome measures and secondary outcome measures at pre-intervention, post-treatment (i.e., 4 weeks after the last intervention session, at the end of the withdrawal phase), and at 6-month follow-up.

DETAILED DESCRIPTION:
Rationale: Patients with post-traumatic stress disorder (PTSD) experience highly frequent and distressing intrusive images depicting earlier aversive experiences. Not only patients with PTSD experience these intrusions; they are also very common in depression. Therefore, trauma treatments that target these intrusions may also benefit patients with depression. Additionally, comorbid depression in patients with PTSD reduces the effects of trauma treatment. It is currently unknown which treatment for traumatic intrusions is most effective for patients who meet criteria for PTSD, depression, or both, and treatment selection is often a process of trial and error. The mechanisms of action of trauma treatments may inform us how to select the most appropriate treatment for a particular individual.

Objective:

The investigators' primary objective is to investigate which treatment (EMDR vs. IR) is most effective for different groups of patients who experience intrusions: patients with PTSD, patients with depression, or patients with PTSD and a comorbid depression. To this end, the investigators will examine the reduction in the severity of intrusions (i.e., frequency, uncontrollability, and degree of interference with daily life). The investigators' secondary objective is to gain more insight into the mechanisms of action of EMDR and IR. To this end, the investigators will examine the role of various mediators of the treatment effects (i.e., the reduction in the severity of intrusions). The investigators will specifically investigate the potential mediating roles of self-compassion, emotion regulation, positive affect, rumination, and the vividness, distress, and associated meaning of intrusions.

Study design: This study will use a single-case experimental design (SCED). In this design, a small group of patients is followed throughout their treatment. It is a within-subjects design in which each patient undergoes a baseline phase (2 weeks prior to the start of treatment) in which no intervention takes place, an experimental phase with treatment interventions (at least 2.5 weeks), and finally a withdrawal phase (4 weeks following the last intervention session) in which no further treatment takes place.

Study population: This study will recruit 42 patients meeting criteria for either PTSD or depression, or for both disorders.

Intervention (if applicable): Patients will be randomly assigned to standard treatments EMDR or IR. In each condition, patients will receive two 75-minute sessions of EMDR or IR each week, as well as an additional coaching session each week. Treatment length depends on patients' needs and varies between 2.5 and 6 weeks.

Main study parameters/endpoints: The primary outcome is a brief measure of characteristics of intrusions (specifically, the frequency, uncontrollability, and degree of interference with daily life), which will be assessed twice daily via an online mobile app.

Additionally, process measures indexing possible mediators concern brief questionnaires on emotion regulation, self-compassion, rumination, positive affect, and the vividness, distress, and related meaning of intrusions, which also serve as the investigators' primary outcome measures. These questionnaires will be assessed daily. All primary outcome measures will be administered during the baseline, experimental, and withdrawal phase. Secondary outcome measures concern questionnaires on quality of life, depression symptoms, and PTSD symptoms which are endorsed at the pre-intervention assessment (i.e., 2 weeks prior to the first intervention session), post-treatment assessment (i.e., 4 weeks after the last intervention session, at the end of the withdrawal phase), and at 6-month follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 70 years
* experiencing intrusions and/or nightmares
* meet criteria for unipolar depressive disorder, PTSD, or both disorders
* past aversive events still cause considerable distress
* be available for trauma treatment twice a week, with an additional coaching session each week
* be proficient in the Dutch language.

Exclusion Criteria:

* the presence of a dissociative identity disorder
* acute suicide risk
* acute psychosis
* substance use disorder
* bipolar disorder type 1 and 2. Other comorbid disorders are allowed.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-01-28 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Severity of intrusions | Severity of intrusions is assessed 2x daily from 2 weeks before treatment up to 1 month after treatment. The severity of intrusions is also assessed 2 weeks prior to the first treatment session, and 1 and 6 months after the last treatment session.
  The severity of intrusions will be computed as a composite score of the frequency, uncontrollability, and degree of interference with daily life. A questionnaire inquiring about the frequency, uncontrollability, and degree of interference with daily life of intrusions over the previous 4 hours will be administered twice daily via an online questionnaire. A time frame of 2 hours is set within which patients are asked to complete the questionnaire to increase reliability. The items are "How many intrusions did you experience over the previous 4 hours?", "To what extent do these intrusions interfere with your daily life?", and "To what extent do you perceive these intrusions as uncontrollable?". The frequency of intrusions is presented as an open-ended question, while uncontrollability and interference with daily life are measured on a 10-point Likert scale.
Anxiety and depression | Anxiety and depression are assessed 2x daily from 2 weeks before treatment up to 1 month after treatment. Anxiety and depression are also assessed 2 weeks prior to the first treatment session, and 1 and 6 months after the last treatment session.
  Anxiety and depression will be assessed twice daily using two items (specifically, "How anxious did you feel over the last couple of hours?" and "How depressed did you feel over the last couple of hours?"), using a 10-point VAS scale with as anchor labels 0: "not at all", and 10: "very extreme".
Emotion regulation | The DERS-18 Strategies subscale (3 items) is assessed daily from 2 weeks before treatment up to 1 month after treatment. The entire DERS-SF is administered 2 weeks prior to the first treatment session, and 1 and 6 months after the last treatment session.
  Emotion regulation is measured by the Difficulties in Emotion Regulation Scale (DERS). A short version has been developed (DERS-SF) and is available in Dutch. Possible scores vary from 18 to 90, with higher scores reflecting greater difficulty with emotion regulation.
Self-compassion | Self-compassion subscale (6 items) is administered daily from 2 weeks before treatment up to 1 month after treatment. The entire SCS-SF is administered 2 weeks prior to the first treatment session, and 1 and 6 months after the last treatment session.
  Self-compassion is measured using a shortened version of the Self-Compassion Scale (i.e., SCS-SF). Possible scores range from 12-60, with higher scores reflecting higher self-compassion, and lower scores reflecting lower self-compassion.
Rumination | Brooding and reflection subscales (5 items) are assessed daily from 2 weeks before treatment up to 1 month after treatment. The entire RRS is administered 2 weeks prior to the first treatment session, and 1 and 6 months after the last treatment session.
  The Ruminative Response Scale (RRS) measures the degree of depressive rumination, or repetitive thinking in response to a low mood. Total scores on the RRS-NL range from 22 to 88, with higher scores reflecting a greater tendency towards ruminative thinking.
Positive affect | Positive affect items (10 items) are assessed daily from 2 weeks before treatment up to 1 month after treatment. The entire PANAS will be assessed 2 weeks prior to the first treatment session, and 1 and 6 months after the last treatment session.
  Positive affect is measured using the Positive Affect scale (10 items) of the Positive and Negative Affect Scale (PANAS). High positive affect refers to the extent to which the person feels positively involved in the environment and experiences positive emotions such as enthusiasm, whereas low positive affect refers to the absence of positive feelings. Total scores for the Positive Affect scale range from 10 to 50, with higher scores reflecting greater positive affect.
Vividness of intrusions | Vividness of intrusions is assessed daily from 2 weeks before treatment up to 1 month after treatment. The vividness of intrusions is also assessed 2 weeks prior to the first treatment session, and 1 and 6 months after the last treatment session.
  The investigators will measure the degree of 'vividness' of intrusions to measure the impact of the interventions. The vividness of intrusions will be measured using an online questionnaire, with the specific item "How vivid are your intrusions right now, on a scale from 0 to 100?", with higher scores reflecting higher vividness.
Distress of intrusions | Distress of intrusions is assessed daily from 2 weeks before treatment up to 1 month after treatment. Additionally, the distress of intrusions is assessed 2 weeks prior to the first treatment session, and 1 and 6 months after the last treatment session.
  The investigators will measure the level of 'distress' of intrusions to measure the impact of the interventions. The distress of intrusions will be measured using an online questionnaire, with the specific item "How distressing are your intrusions right now, on a scale from 0 to 100?", with higher scores reflecting higher distress.
Intrusion-related beliefs | Intrusion-related beliefs are assessed 2 weeks prior to the first treatment session, and 1 and 6 months after the last treatment session.
  The investigators will assess the content and believability of 'intrusion-related beliefs about oneself', in order to measure the change in the meanings associated with the intrusions. This outcome measure will be assessed using an online questionnaire, with the specific items "What do your intrusions say about you?" (open ended question), and "How believable is this belief right now, on a scale from 0 to 100?", with higher scores reflecting stronger intrusion-related beliefs about oneself.

SECONDARY OUTCOMES:
The Posttraumatic Stress Disorder Checklist for DSM-5 | The PCL-5 will be administered 2 weeks prior to the first treatment session, and 1 and 6 months after the last treatment session.
  The Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5) is a 20-item self-report questionnaire that measures the severity of PTSD symptoms in the past month. The PCL-5 contains four subscales: Intrusions (items 1-5), Avoidance (items 6-7), Negative Change in Cognitions and Mood (NACM; items 8-14), and Change in Arousal and Reactivity (AR; items 15-20).
The Beck Depression Inventory II | The BDI-II will be administered 2 weeks prior to the first treatment session, and 1 and 6 months after the last treatment session.
  The Beck Depression Inventory II (BDI-II) is a 21-item self-report questionnaire that measures the severity of depressive symptoms over the past 2 weeks. Possible scores range from 21 to 63, with higher scores reflecting more severe depressive symptoms.
Mental Health Quality of Life 7D | The MHQoL will be administered 2 weeks prior to the first treatment session, and 1 and 6 months after the last treatment session.
  The Dutch version of the Mental Health Quality of Life 7D (MHQoL) measures quality of life in people with mental health problems. The instrument consists of 7 self-report items in the domains of self-image, independence, mood, relationships, daily activities, physical health, and future. Possible scores range from 0 to 21, with higher scores reflecting a higher quality of life.
The Credibility/Expectancy Questionnaire | The CEQ is assessed twice weekly from 2 weeks before treatment up to 1 month after treatment. The CEQ is also assessed 2 weeks prior to the first treatment session, and 1 and 6 months after the last treatment session.
  The Credibility/Expectancy Questionnaire (CEQ) is a questionnaire that consists of six questions: four questions considering the treatment credibility, and two questions considering treatment expectancy.

OTHER OUTCOMES:
MINI Neuropsychiatric Interview | The MINI Interview will be administered at the pre-intervention assessment (2 weeks prior to the first treatment session) to determine whether a patient meets the inclusion criteria and to describe other comorbidities in the sample.
  The MINI Neuropsychiatric Interview (MINI-S for DSM-5 version) is a structured diagnostic interview that will be used to screen for mental health diagnoses (i.e., both inclusion and exclusion criteria).
Life Events Checklist for the DSM-5 | The LEC-5 will be administered at the pre-intervention assessment (2 weeks prior to the first treatment session).
  The purpose of the administration of the LEC-5 is to gather information about potentially traumatic experiences that patients may have experienced. The LEC-5 does not have an official scoring protocol or interpretation of scores. Rather, it is used to identify whether a patient has experienced a traumatic event.

CONTACTS AND LOCATIONS:
Locations (1):
- Geestelijke Gezondheidszorg Eindhoven, Eindhoven, North Brabant, Netherlands

REFERENCES:
- [Background] Arntz A, Weertman A. Treatment of childhood memories: theory and practice. Behav Res Ther. 1999 Aug;37(8):715-40. doi: 10.1016/s0005-7967(98)00173-9. PMID 10452174
- [Background] Beck, A. T., Steer, R., Brown, G. (1996). Manual for the Beck Depression Inventory-II. San Antonio: The Psychological Corporation.
- [Background] Boeschoten, M.A., Bakker, A., Jongedijk, R.A., & Olff, M. (2014). PTSD Checklist for DSM-5-Nederlandstalige versie. Uitgave: Stichting Centrum '45, Arq Psychotrauma Expert Groep, Diemen
- [Background] De Jongh, A., & Ten Broeke, E. (2013). Handboek EMDR: Een geprotocolleerde behandelmethode voor de gevolgen van psychotrauma [EMDR manual: A protocolised treatment method for the consequences of psychotrauma]. Amsterdam: Pearson Assessment and Information B.V.
- [Background] Gratz, K. L., & Roemer, L. (2004). Multidimensional assessment of emotion regulation and dysregulation: Development, factor structure, and initial validation of the difficulties in emotion regulation scale. Journal of Psychopathology and Behavioral Assessment, 26(1), 41-54. https://doi.org/10.1023/B:JOBA.0000007455.08539.94
- [Background] Kaufman EA, Xia M, Fosco G, Yaptangco M, Skidmore CR, Crowell SE. The Difficulties in Emotion Regulation Scale Short Form (DERS-SF): Validation and Replication in Adolescent and Adult Samples. J Psychopathol Behav Assess. 2016 Sep;38(3):443-455. doi: 10.1007/s10862-015-9529-3. Epub 2015 Nov 23. PMID 41522882
- [Background] Amorim P, Lecrubier Y, Weiller E, Hergueta T, Sheehan D. DSM-IH-R Psychotic Disorders: procedural validity of the Mini International Neuropsychiatric Interview (MINI). Concordance and causes for discordance with the CIDI. Eur Psychiatry. 1998;13(1):26-34. doi: 10.1016/S0924-9338(97)86748-X. PMID 19698595
- [Background] Neff, K. D. (2003). The development and validation of a scale to measure self-compassion. Self and Identity, 2(3), 223-250. https://doi.org/10.1080/15298860309027
- [Background] Neff KD, Vonk R. Self-compassion versus global self-esteem: two different ways of relating to oneself. J Pers. 2009 Feb;77(1):23-50. doi: 10.1111/j.1467-6494.2008.00537.x. Epub 2008 Nov 28. PMID 19076996
- [Background] Neumann A, van Lier PA, Gratz KL, Koot HM. Multidimensional assessment of emotion regulation difficulties in adolescents using the Difficulties in Emotion Regulation Scale. Assessment. 2010 Mar;17(1):138-49. doi: 10.1177/1073191109349579. Epub 2009 Nov 14. PMID 19915198
- [Background] Nolen-Hoeksema S, Morrow J. A prospective study of depression and posttraumatic stress symptoms after a natural disaster: the 1989 Loma Prieta Earthquake. J Pers Soc Psychol. 1991 Jul;61(1):115-21. doi: 10.1037//0022-3514.61.1.115. PMID 1890582
- [Background] Overbeek, T., & Schruers, K. (2019). Mini International Neuropsychiatric Interview - Simplified (MINIS) voor DSM-5, Nederlandse versie.
- [Background] Raes, F. (2009). Ruminative Response Scale--Revised; Dutch Version (RRS-NL, RRS) [Database record]. APA PsycTests. https://doi.org/10.1037/t66234-000
- [Background] Raes F, Pommier E, Neff KD, Van Gucht D. Construction and factorial validation of a short form of the Self-Compassion Scale. Clin Psychol Psychother. 2011 May-Jun;18(3):250-5. doi: 10.1002/cpp.702. Epub 2010 Jun 8. PMID 21584907
- [Background] Shapiro F. (2001). Eye movement desensitization and reprocessing (EMDR): basic principles, protocols and procedures. 2nd ed. New York, NY: The Guilford Press.
- [Background] Topper M, Emmelkamp PM, Watkins E, Ehring T. Development and assessment of brief versions of the Penn State Worry Questionnaire and the Ruminative Response Scale. Br J Clin Psychol. 2014 Nov;53(4):402-21. doi: 10.1111/bjc.12052. Epub 2014 May 2. PMID 24799256
- [Background] van Krugten FC, Kaddouri M, Goorden M, van Balkom AJ, Bockting CL, Peeters FP, Hakkaart-van Roijen L; Decision Tool Unipolar Depression (DTUD) Consortium. Indicators of patients with major depressive disorder in need of highly specialized care: A systematic review. PLoS One. 2017 Feb 8;12(2):e0171659. doi: 10.1371/journal.pone.0171659. eCollection 2017. PMID 28178306
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Weathers, F.W., Litz, B. T., Keane, T. M., Palmieri, P. A., Marx, B. P., & Schnurr, P. P. (2013). The PTSD Checklist for DSM-5 (PCL-5). Retrieved on December 1, 2023 from https://www.ptsd.va.gov/professional/assessment/adult-sr/ptsd-checklist.asp#obtai